CLINICAL TRIAL: NCT01949064
Title: Anwendung Von Elektromyographie Mit Gleichzeitigem Bio-Feedback Zur Behandlung Von Craniomandibulären Dysfunktionen Und/Oder Bruxismus.
Brief Title: Use of Electromyography With Bio-Feedback for the Treatment of Craniomandibular Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Giannakopoulos Nikolaos, Dr.med.dent., M.Sc., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BioGC1UHeidelberg
Record Dates: First submitted 2013-09-17; First posted 2013-09-24 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Craniomandibular Dysfunction; Orofacial Pain
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Michigan-type occlusal splint (Active Comparator): Occlusal splint, Michigan-type
  Interventions: Device: Michigan-type occlusal splint
- Grindcare (Active Comparator): Biofeedback device
  Interventions: Device: Grindcare

INTERVENTIONS:
Device: Grindcare
  Arms: Grindcare
Device: Michigan-type occlusal splint
  Arms: Michigan-type occlusal splint

SUMMARY:
The treatment of craniomandibular disorders is a challenging task. Many different treatments are yet available with occlusal splints being one of the most commonly used. A relative new diagnostic and treatment alternative is the Grindcare device. This enables the electromyographic (EMG) assessment of the activity of the temporal muscle and the contigent electrical stimulation of this muscle as bio-feedback whenever the EMG activity exceeds a certain limit. This stimulation results to a sudden break of the muscle activity.

Aim of this study is to compare the therapeutic efficacy of the Grindcare device in pain reduction at female non-chronic CMD patients to that of a Michigan-type splint. Our null-hypothesis was that there is no difference between the device and the splint in the reduction of pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age between 18 and 70 years
* Non-chronic painful CMD with/without mandibular movement restriction
* Female

Exclusion Criteria:

* Pregnancy or breastfeeding
* Chronic Pain Status higher than 2
* Known allergic reaction against the gel pads
* Electronic implants (pacemaker, defibrilator, insulin pump)
* Facial pain of dental or neuropathic etiology
* Traumatic injuries of the face / operations
* Dental treatment need
* Problems with swallowing reflex

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Worst perceived pain | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Nikitas Giannakopoulos, Dr.med.dent,M.Sc, Principal Investigator — Poliklinik für Zahnärztliche Prothetik
Locations (1):
- Poliklinik für Zahnärztliche Prothetik, Heidelberg, Germany